CLINICAL TRIAL: NCT02086643
Title: The Retroclavicular Approach for Regional Anesthesia of the Upper Limb in Patients With BMI ≥ 30 kg/m2 : A Descriptive Study
Brief Title: The Retroclavicular Approach for Regional Anesthesia of the Upper Limb in Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Pablo Echave, Anesthesiologist, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-175
Record Dates: First submitted 2014-03-08; First posted 2014-03-13 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Overweight
Keywords: Infraclavicular block; Brachial Plexus; Retroclavicular Approach; Complications of retroclavicular approach; Success of retroclavicular approach; Obese Patients; Obesity and Anesthesia
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retroclavicular block (Experimental): Retroclavicular block
  Interventions: Procedure: Retroclavicular block

INTERVENTIONS:
Procedure: Retroclavicular block — Retroclavicular ultrasound guided nerve block with total injection of 40 ml of a mixture of 20 ml ropivacaine 0,5% (5 mg/ml) + 20 ml mepivacaine 1,5% (15 mg/ml) + epinephrine 1 : 400 000 (2,5 mcg/ml). Incremental injections of 5 ml separated by an aspiration test.

SUMMARY:
The goal of this study is to determine the success rate of the retroclavicular approach for the anesthesia of the upper limb in the obese patient population (BMI ≥ 30 kg/m2)

DETAILED DESCRIPTION:
Classic infraclavicular approach of the brachial plexus involves a needle puncture below the clavicle and advancing the needle with a 45-60 degree angle from cephalad to caudad. The aim is to advanced the block needle posterior to the axillary artery and to deposit the local anesthetic at that point, near the posterior cord. A "U" shaped spread around the artery should ensure distribution around all three cords. Ultrasound guidance is highly recommended and neurostimulation is optional.

The retroclavicular approach is a variant to this classical technique. Ultrasound probe is positioned initially below the clavicle in a manner similar to the classic approach but is then rotated in a clockwise fashion (right arm) or counter-clockwise fashion (left arm) for about 25-35 degrees. The puncture site is just behind the clavicle at the most lateral point available. If initial entry point is optimal, needle direction is then parallel to ultrasound probe. The final aim and position of block needle is identical to classical approach. Entry point ensures a parallel alignment of the needle and the ultrasound beam, thus enabling almost perfect visualization of both artery, cords and block needle. This is turn optimizes safety, rapidity of technique, efficiency and efficacy.

It is recognized that regional anesthesia is more difficult to perform in obese patients. Anatomic landmarks are harder to localize in this population and ultrasound guidance is more difficult because of the attenuation of the ultrasound beam by adipose tissue. The complication rate of regional techniques is also reported to be higher in the obese patient population.

Since the retroclavicular variant of the infraclavicular approach for the anesthesia of the brachial plexus offers a better needle visualisation, we believe that this technique can be used successfully in the obese patient population with a low complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Elective or Urgent Surgery of the hand, wrist or forearm
* 18 years and older
* Ability to consent
* American Society of Anesthesiologists class 1 to 3
* BMI ≥ 30 kg/m2

Exclusion Criteria:

* Infection at the site of infection
* Abnormal anatomy at the site of infection
* Coagulopathy
* Severe Pulmonary Disease
* Preexisting neurological symptom(s) in the operated arm
* Pregnant patients
* Patients weighing less than 50 kg
* Allergy to amide type local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Surgery completion under regional block | Success is defined at end of surgery for which block was done, generally within 1 to 3 hours after block is performed
  Success rate is defined as the completion of the intended surgery under regional anesthesia with retroclavicular block without the need for a rescue technique. These techniques are defined as: adding local anesthetic locally by surgeon, rescue intravenous narcotics in excess of 1 microgram per kilogram of patient weight, need for general anesthesia, rescue distal neural blockage by anesthesiologist. Patient sedation with midazolam 1 to 2 mg IV or propofol perfusion up to 50 mcg/kg/min is allowed for patient comfort during the surgery and is not considered a rescue technique.

SECONDARY OUTCOMES:
Sensitive block progression | Assessed 10, 20 and 30 minutes after block completion
  Progress of the sensory block in the distribution of the radial, median, ulnar, musculocutaneous, and medial cutaneous nerves of the forearm and hand at 10, 20 and 30 minutes after block completion (mepivacaine-ropivacaine mixed injection). The scale used is: 0:no sensitive block, 1:analgesia (loss of pain but not tactile sensation), 2:anesthesia (loss of pain and tactile sensation).
Motor Block Progression | Assessed 10, 20, 30 minutes after the block
  Progress of the motor block in the distribution of the radial, median, ulnar, musculocutaneous nerves of the forearm and hand at 10, 20, and 30 minutes after block completion (mepivacaine injection). The scale used is: 0: no motor block, 1: paresis, 2: paralysis. No units are attached to this scale
Technique duration | Time required in seconds for the retroclavicular block technique completion, generally under 15 minutes
  Number of seconds needed to complete the block, from time of local skin anesthesia until regional block needle removal (local skin anesthesia plus injection of mepivacaine-ropivacaine mixture)
Needle visualization | Assessed after study completion, once all 30 patients will have been completed. Assessment will take place in the first 4 weeks after all 30 patients have been recruited
  Using the Likert standardized scale, two evaluators will individually quantify the ease of needle visualization using the video footage recorded by the ultrasound machine from all the retroclavicular blocks. Likert scale for visualization, is defined as: 1:very bad, 2: bad, 3: adequate, 4:good, 5: very good.
Patient discomfort | Assessed 1 minute after block completion
  Using a Visual Analog Scale (VAS), patients will quantify the discomfort they experienced during the block. This assessment will take place in the minutes following mepivacaine injection and block needle withdrawal. The VAS scale is rated from 1-10, 1 being almost no pain and 10 being the worst pain ever.
Patient satisfaction | Assessed 48 hours after the block
  Using a VAS, patients will quantify their satisfaction with the retroclavicular technique throughout the study period.
Late Complication Rate | Assessed 48 hours after the block
  With a phone call to the patient at 48 hours after injection of mepivacaine-ropivacaine mixture, complications will be searched for (pain at puncture site, paresthesia or paresis in the operated arm, signs of infection at puncture site such as redness or purulent discharge). Response is classified as YES or NO. No units attached to this scale. If patient reports paresthesia or paresis, further questioning over the phone will determine which nerve or cord is involved.
Duration of the Block's Effects | Assessed 48 hours after the block
  Duration of the block will be evaluated using 3 criteria: patient's subjective opinion of when the block receded (time of the day), time at which first oral analgesia is taken, and time of first onset of pain. Units involved is time (for example "3 pm".)
Use of narcotic for tourniquet pain | Assessed while surgery in under process
  If at any point during the surgery, patient complains of tourniquet pain, this will be noted as well as the analgesia given. Units is time of pain ("3 pm") and analgesia given ("micrograms of fentanyl").
Rate of Neurostimulation Usage | Assessed during the block
  At the discretion of the anesthesiologist performing the block, neurostimulation can be used to supplement ultrasound guidance. This will be recorded as a YES or NO (neurostimulation used or not). No units attached to this rate.
Failure because of poor ultrasound visualization | Assessed during the performance of the nerve block
  If, for a given patient, during ultrasound guidance the anatomic structure are too poorly visualized to safely perform the block, no puncture will be attempted and the technique will be considered a failure; an alternative anesthesia technique will be proposed to the patient.
Early Complication Rate | Assessed during block performance, throughout surgery and in the PACU. Generally during a period of 4-6 hours after block completion
  Immediate and early complications (vascular puncture, pneumothorax, paresthesia during block performance, pain during infection of the local anesthetics, Horner's syndrome) will be assessed throughout the patient's stay in the OR and PACU. Immediate and appropriate treatment will be provided if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Echave, M.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec, Canada